CLINICAL TRIAL: NCT03150147
Title: A Randomized Controlled Trial Comparing Non-ischemic Hypothermic Cardioplegic Perfusion to Ischemic Cold Static Preservation of Donor Hearts in Adult Cardiac Transplantation
Brief Title: A Randomized Controlled Trial Comparing Non-ischemic to Ischemic Preservation in Adult Cardiac Transplantation
Acronym: NIHP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Johan Nilsson, MD, PhD, Professor, Region Skane
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2016/603
Record Dates: First submitted 2017-05-08; First posted 2017-05-12 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Transplant; Failure, Heart
Keywords: Organ preservation; Survival; Graft function; Reperfusion injury; Heart transplantation
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Intervention Model Description: Initially the study is a single center, prospective, open, blinded endpoint, non-randomized, controlled clinical trial. Six patients will be transplanted with the NICHCP method. These will be compared with contemporary control patients transplanted with standard ICSS (N=25). An analyze will be performed when these six patients has passed 180-days post-transplant. The result will be reported.
  After the the initially study has been completed, the study will become a single center, prospective, open, blinded endpoint, randomized, controlled clinical trial. The continued study will comprise 17 patients in the test group and 17 control patients. The main outcomes will be reported on intention to treat basis. PGD and ACR assessment will be performed by a blinded access. Randomisation will be computer generated.
Who Masked: Participant, Outcomes Assessor
Masking Description: PGD and ACR assessment will be performed by a blinded access
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-ischemic preservation. (Experimental): Non-ischemic hypothermic perfusion (NIHP): The device, a portable heart-lung machine, is continous/intermittent perfused the heart with a new preservation solution at a temperature of 8°C.
  Interventions: Other: Non-ischemic preservation
- Standard ischemic storage. (Other): Ischemic cold static storage: a crystalloid solution (cardioplegia) is used to stop and preserve the heart. The heart is storage i a transport box containing ice to keep the temperature around 8°C.
  Interventions: Other: Ischemic cold static storage

INTERVENTIONS:
Other: Non-ischemic preservation — The device is a portable heart-lung machine; an automatic pressure and flow-controlled perfusion system. The heart is submerged in a solution and the medium is circulated in the heart, at a temperature of 8°C.
  Arms: Non-ischemic preservation.
Other: Ischemic cold static storage — Standard ischemic cold static storage; a crystalloid solution (cardioplegia) is used to stop and preserve the heart. Cardioplegia is given. The heart is storage i a transport box containing ice to keep the temperature around 8°C.
  Arms: Standard ischemic storage.

SUMMARY:
The overall aim of this proposal is to compare a new state-of-the-art ex-vivo organ preservation method with standard ischemic cold static storage of donor hearts in adult cardiac transplantation.

Standard heart preservation before transplantation consists of cold ischemic storage of the heart. Clinical studies has shown that the morbidity and mortality risk increases with extension of the allograft ischemic time over four hours. For each additional hour the mortality risk increase with 25% the first year. This time constrained is costly and results in severe logistical problems, leading to loss of transplantable organs.

Initially the study is prospective, single-institution, open-label, non-randomised trial comparing the NIHP method with the conventionally SCS in adult heart transplanted patients at Skane University Hospital, Lund, Sweden. Six patients will be transplanted using the non-ischemic hypothermic cardioplegic perfusion. These will be compared with contemporary control patients transplanted with standard ischemic cold static storage. The results will be analysed and reported.

After the initially six patients have been completed, the study will become a single center, prospective, open, blinded endpoint, randomized, controlled clinical trial including 34 patients.

The primary end-point is a composite of mortality, primary graft dysfunction (PGD), need for extra corporal support, or acute cellular rejection (ACR) within 30- days post-transplant. PGD and ACR will be accessed blinded.An improved preservation of the transplanted organ will reduce the major limitations for survival in the early post-transplant period such as non-specific graft failure and acute rejection. Furthermore, it will make it possible to increase the donor pool.

DETAILED DESCRIPTION:
SURVEY OF THE FIELD

Ischemia and reperfusion (I/R)-elicited tissue injury contributes to morbidity and mortality4. In organ transplantation, it is a major challenge. The imbalance in metabolic supply and demand within the ischemic organ results in tissue hypoxia and microvascular dysfunction4. The following reperfusion enhances the activation of innate and adaptive immune responses resulting in a cell death programs4,5. Furthermore, it has been report that miRNA expression profile for heart transplantation is associated with I/R injury. Standard heart preservation before transplantation consists of cold ischemic storage of the heart. Clinical studies have shown that the mortality risk increases sharply with extension of the allograft ischemic time over 4 hours. For each additional hour, the mortality risk increase with 25% the first year. Different myocardial cardioplegic preservation solutions and an ex-vivo perfusion machine have been developed. That technique includes use of whole blood from deceased donor and a normothermic beating heart consuming nutrients during the preservation. Despite some promising experimental results, no consistent differences in outcome have been found. Improved preservation of the endothelium of the coronary arteries is instrumental to achieve improved patient short and long term outcome. A damaged endothelium could result in cardiac allograft vasculopathy (CAV) and increases the risk of ACR. Therefore, prolonged time and improved storage of the donor heart would save lives.

PURPOSE AND AIM

The overall aim of this study is to compare a new state-of-the-art organ preservation technique, non-ischemic continous/intermittent hypothermic cardioplegic perfusion (NICHCP), on immediate and long term heart allograft function and rejection episodes, with standard ischemic cold static storage (ICSS) of donor hearts in adult cardiac transplantation.

A new ex-vivo heart perfusion technique where the heart is perfused during explantation, using an independent portable heart-lung-machine, has been developed by Prof. Steen's research group3. Pre-clinical studies have shown that the new technology using NICHCP of donor hearts can be safely applied for 24 hours in pigs, however this new perfusion technique has never been used on man.

The primary hypothesis is that the NICHCP is superior to ischemic cold static storage of donor hearts. The primary end-point is a composite of mortality, primary graft dysfunction, need for extra corporal mechanical support, or Acute Cellular Rejection (ACR) ≥ grade 2 within 30-days.

RESEARCH QUESTION

The study will investigate the superiority of the new methodology (NICHCP) in terms of improved immediate and prolonged organ function. More specifically, it is hypothesized that the weaning period of cardio-pulmonary bypass, will be shorter, the need for inotropic support reduced, and the major limitations for survival in the early post-transplant period such as non-specific graft failure, multiorgan failure, ACR, and infection will decrease. Furthermore, in the late post-transplant period, it is hypothesized that the development of CAV and immunosuppressive side effects, such as malignancy, will be reduced.

WORK PLAN

In the initial phase, it is excepted that 1 - 2 patients will be enrolled per month. During the randomized part of the study It is expected to enroll 1 - 4 patients per month. With that pace, the study is completed within about 24 months. The patient short term follow-up is 30 days and long term follow up is 12 months. For short-term-analysis purpose the study is considered completed as the last patient of the study has passed 30-days post-surgery. The long-term study will continue to monitor the patients for 12 months. Adverse events will be recorded even if occurring after completion of the study and all patients will be followed throughout life according to standard clinical care.

If this is successful, this will be introduced as standard among other national and international collaborators. The investigators estimate that this technique will be the golden standard within 5 years.

STUDY DESIGN

Initially the study is a prospective, single-institution, open-label, non-randomised trial. Here, six patients will be transplanted with the NICHCP method. These will be compared with contemporary control patients transplanted with standard ICSS. An interim assessment will be performed when these six patients has passed 180-days post-transplant. The results from this study will be analysed and published. A report will be sent to the Ethical review bord for an approval to continue with the second part of the study.

After six patients have been transplanted with the NICHCP method and a new approval has been achieved from the local ethical board, the study will become a single center, prospective, open, blinded endpoint, randomized, controlled clinical trial. The continued study will comprise 17 patients in the test group and 17 control patients. The main outcomes will be reported on intention to treat basis. PGD and ACR assessment will be performed by a blinded access. Listed heart recipients (aged >18 years) at Skåne University Hospital will be screened. Patients who full-fill all inclusion and no exclusion criteria will be included after they signed the informed consent form. In the initial phase, it is excepted that 1-2 patients will be enrolled per month. During the randomized part of the study it is expected to enroll 1-4 patients per month. With that pace, the study is completed within 24 months. The patient short term follow-up is 30 days and long term follow up is 12 months. For short-term-analysis purpose the study is considered completed as the last patient of the study has passed 30-days post-surgery. The long-term study will continue to monitor the patients for 12 months. Adverse events will be recorded even if occurring after completion of the study and all patients will be followed throughout life according to standard clinical care.

STATISTICAL ANALYS PLAN

Descriptive statistics will be presented as means, standard deviations, medians and inter quartile ranges for the continuous variables and as counts and percent for categorical variables. An alpha level of 5% will be used for all analyses, unless otherwise stated. Demographics will be tabulated overall and by treatment group. The results from the laboratory analysis will be calculated based on continuous variables. All data analyses will be performed on data available. After three of the patients have been enrolled a safety assessment will be performed. An interim assessment of the initial six patients in the test group will be performed when all six patients has passed 30-days post-transplant or expired. A protocol deviation is any event where investigator or study personnel did not conduct the study per the protocol or applicable laws. All deviations will be reported to the Principal Investigator (regardless of cause or prior approval) and will be noted on the eCRF form.

CLINICAL AND SCIENTIFIC IMPLICATIONS

The use of an ex-vivo machine for the preservation of a donor heart requires more resources than the technology used today, such as special equipment, suitable transportation and bank blood to prime the perfusion module. Compared with cold static techniques for preservation, this will initially be costly. However, this must be weighed against the value of more donor hearts become available for transplant and cost savings in the form of shorter time to perform the surgery, reduced incidence of the primary graft dysfunction (PGD), less need for expensive mechanical cardiac support post-transplant, shortened hospitalization and longer-term risk reduction of chronic rejection. The costs of complications directly connected to the transplant is cost driven, especially if the recipient develops PGD requiring mechanical circulatory support with a prolonged ICU stay. Furthermore, in the future the transplantation can be scheduled to day-time surgery and complexed high risk cases can be done with the highest competence available without time limitation. An improved preservation of the transplanted organ will reduce the major limitations for survival in the early post-transplant period such as PGD. Furthermore, it will make it possible to increase the donor pool. Theoretically in the nordic countries, this would enable international organ sharing with Europe and the eastern United States. This expansion of the donor pool is one of the main potential benefits of this device.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Listed for heart transplantation
* Signed informed consent form

Exclusion Criteria:

* Previous solid organ or bone marrow transplantation
* 4 or more previous sternotomies
* known malignancy
* kidney failure (estimated creatinine clearness, GFR <30)
* liver failure (ASAT, ALAT or total Bilirubin) > 5 times upper limit of normal, or INR >2.0,
* ongoing septicemia
* systemic inflammatory disorders treated with corticosteroids
* not able to understand Swedish

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Short-term graft failure | Within 30-days post-transplantation
  The Primary End-Point is defined as a composite endpoint of patient death due to graft failure, re-transplantation due to graft failure, severe primary graft dysfunction (PGD), need for extra corporal mechanical support such as ECMO within 7 days post transplantation, or acute cellular rejection (ACR) ≥ grade 2.
  PGD grading is done according to the International Society of Heart and Lung Transplantation guidelines. ACR assessment is based on post-transplant myocardial biopsy information and standard clinical evaluation.

SECONDARY OUTCOMES:
Long-term graft failure | Within 12-months post-transplantation
  Secondary End-Points is defined as a time to the composite endpoint defined as: severe primary graft dysfunction (PGD), need for extra corporal mechanical support such as ECMO, acute cellular rejection (ACR) ≥ grade 2, or CAV.
  CAV assessment is based on information from the angiography and registered according to the International Society of Heart and Lung Transplantation guidelines guidelines. ACR assessment is based on post-transplant myocardial biopsy information and standard clinical evaluation.
Ischemia and reperfusion injury | Within 30-days post-transplantation
  CK-MB are measured from blood samples that are collected from the sinus coronaries after finalized preservation, and from blood-samples 6, 12, 24, 48, and 72 hours after release of x-clamp.
Ischemia and reperfusion injury | Within 30-days post-transplantation
  cTnl are measured from blood samples that are collected from the sinus coronaries after finalized preservation, and from blood-samples 6, 12, 24, 48, and 72 hours after release of x-clamp.

OTHER OUTCOMES:
Postoperative renal function | Within 30-days post-transplantation
  The renal function is analyzed based on s-Creatinine levels, need for dialysis (days).
Postoperative liver function | Within 30-days post-transplantation
  The liver function is measured with ASAT and ALAT.
Length of Stay | Within 12-months post-transplantation
  Intensive Care Unit (ICU): Calculated from time patient arrives into the ICU until the patient is discharged from the ICU. Hospital: Calculated from date and time of surgery until date and time that the patient is discharged from the hospital.
EQ-5D | Within 12-months post-transplantation
  The EuroQol (EQ-5D) is an instrument used to assess the current health status of patients. It consists of five domains and one visual analogue scale. This instrument assesses morbidity, self-care, usual activity, pain, and anxiety and depression of patients. The EQ-5D will be completed at 1, 3, 6, and 12 months visits.
Immediate Cardiac function - weaning time | Within 2-days post-transplantation
  The immediate organ function is determined as the time for weaning off cardiopulmonary bypass (CPB) measured in minutes.
Organ graft dysfunction due to rejection | Within 12-months post-transplantation
  Patient death due to graft failure, re-transplantation or sign of graft rejection (ACR ≥ grade 1, AMR ≥1 or CAV) after transplantation. ACR assessment is based on post-transplant myocardial biopsy information and standard clinical evaluation
Organ preservation injury | Within 1-days post-transplantation
  Measure of IL-1, IL-6, TNF, micro-RNAs in tissue samples taken from the donor heart
Immediate Cardiac function - inotropic support score | Within 48-hours post transplantation
  Summarize of inotropic support according to the definition in the PGD grading, International Society of Heart and Lung Transplantation guidelines.
Respiratory dysfunction | Within 7 days post-transplantation
  Need for re-intubation or time on ventilator > 48 hours
Organ rejection | Within 12-months post-transplantation
  Measure of donor specific cell free DNA each month post transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Johan Nilsson, MD, PhD, Principal Investigator — Lund University and Skåne University Hospital
Locations (1):
- Skane University Hospital, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nilsson J, Ohlsson M, Hoglund P, Ekmehag B, Koul B, Andersson B. The International Heart Transplant Survival Algorithm (IHTSA): a new model to improve organ sharing and survival. PLoS One. 2015 Mar 11;10(3):e0118644. doi: 10.1371/journal.pone.0118644. eCollection 2015. PMID 25760647
- [Background] Messer S, Ardehali A, Tsui S. Normothermic donor heart perfusion: current clinical experience and the future. Transpl Int. 2015 Jun;28(6):634-42. doi: 10.1111/tri.12361. Epub 2014 Jul 7. PMID 24853906
- [Background] Steen S, Paskevicius A, Liao Q, Sjoberg T. Safe orthotopic transplantation of hearts harvested 24 hours after brain death and preserved for 24 hours. Scand Cardiovasc J. 2016 Jun;50(3):193-200. doi: 10.3109/14017431.2016.1154598. Epub 2016 Apr 4. PMID 26882241
- [Background] Jernryd V, Metzsch C, Andersson B, Nilsson J. Organ Preservation and Reperfusion Influence on Outcome after Heart Transplantation. The Journal of Heart and Lung Transplantation , Volume 35 , Issue 4 , S193
- [Background] Zhou L, Zang G, Zhang G, Wang H, Zhang X, Johnston N, Min W, Luke P, Jevnikar A, Haig A, Zheng X. MicroRNA and mRNA signatures in ischemia reperfusion injury in heart transplantation. PLoS One. 2013 Nov 20;8(11):e79805. doi: 10.1371/journal.pone.0079805. eCollection 2013. PMID 24278182
- [Background] Ardehali A, Esmailian F, Deng M, Soltesz E, Hsich E, Naka Y, Mancini D, Camacho M, Zucker M, Leprince P, Padera R, Kobashigawa J; PROCEED II trial investigators. Ex-vivo perfusion of donor hearts for human heart transplantation (PROCEED II): a prospective, open-label, multicentre, randomised non-inferiority trial. Lancet. 2015 Jun 27;385(9987):2577-84. doi: 10.1016/S0140-6736(15)60261-6. Epub 2015 Apr 14. PMID 25888086
- [Background] Qin G, Sjoberg T, Liao Q, Sun X, Steen S. Intact endothelial and contractile function of coronary artery after 8 hours of heart preservation. Scand Cardiovasc J. 2016 Oct-Dec;50(5-6):362-366. doi: 10.1080/14017431.2016.1213876. Epub 2016 Aug 3. PMID 27420646
- [Background] Eltzschig HK, Eckle T. Ischemia and reperfusion--from mechanism to translation. Nat Med. 2011 Nov 7;17(11):1391-401. doi: 10.1038/nm.2507. PMID 22064429
- [Result] Nilsson J, Jernryd V, Qin G, Paskevicius A, Metzsch C, Sjoberg T, Steen S. A nonrandomized open-label phase 2 trial of nonischemic heart preservation for human heart transplantation. Nat Commun. 2020 Jun 12;11(1):2976. doi: 10.1038/s41467-020-16782-9. PMID 32532991